CLINICAL TRIAL: NCT04361578
Title: Prediction of Short-term Outcome in Patients With Acute Closed Traumatic Brain Injury Using Magnetic Resonance Elastography
Brief Title: Magnetic Resonance Elastography in Patients With Acute Closed Traumatic Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, SWLJF, Director, department of Neurotrauma, Xiangya Hospital of Central South University
Other Study IDs: TBI_MRE
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; magnetic resonance elastography; brain compliance
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: All patients enrolled in the study will be in this group.
  Interventions: Diagnostic Test: Magnetic resonance elastography

INTERVENTIONS:
Diagnostic Test: Magnetic resonance elastography — All patients enrolled will receive magnetic resonance elastography of the brain.

SUMMARY:
Traumatic brain injury (TBI) is a major public health issue, and intracranial hypertension in the acute phase remains a critical scientific issue. Many patients with acute closed TBI received conservative, non-surgical treatments at first, while 5%~19% of which develops intractable intracranial hypertension that requires emergent surgery. Therefore, it is of great clinical significance to identify patients who are at high risk of deterioration in the early stage. Previous studies have found that brain compliance is a contributive factor to intracranial pressure, and might serve in the development of intracranial hypertension after TBI. We made assumption that intracranial pressure has a negative relationship with brain compliance providing that the volume of hematoma remains constant. However, few studies have applied magnetic resonance elastography (MRE) in evaluating brain compliance in patients with TBI. Therefore, this study is designed to enroll patients with acute closed traumatic brain injury who are initially treated non-surgically. Magnetic resonance elastography (MRE) sequences are performed to non-invasively assess patients' brain compliances, in the hope of exploring the potential value of MRE biomarkers to predict the short-term outcome in patients with acute closed TBI who are initially receive non-surgical treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old
* Acute closed traumatic brain injury within 7 days
* Not receiving surgical intervention according to the judgement of neurosurgeons
* Expected tolerance of magnetic resonance imaging (MRI) scan 7 days from injury

Exclusion Criteria:

* Vital organ failure: congestive heart failure, respiratory failure, renal failure (CKD≥stage 3), severe hepatic dysfunction (Child-Pugh stage B or C)
* Any central nervous system (CNS) pathology prior to injury: stroke, epilepsy, CNS tumour/infections, dementia or other neurodegenerative diseases
* CT reveals infratentorial hematoma
* Contraindications of MRI
* Currently enrolled in other researches

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with acute closed traumatic brain injury within 7 days will be enrolled in the study. Patients are conservatively managed (didn't receive surgery yet) according to the judgement of neurosurgeons.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
14-day ΔGCS | 14 days after injury
  Change of Glasgow Coma Scale (GCS) 14 days after injury from GCS at admission. The GCS is a indication of patient's conscious status, ranging from 3 (poor) to 15 (good).

SECONDARY OUTCOMES:
14-day mortality | 14 days after injury
  All-cause mortality within 14 days from injury.
14-day emergent surgery | 14 days after injury
  Emergent surgery due to intracranial pathology within 14 days from injury. The decision of emergent surgery (evacuation of newly emerged hematoma, decompressive craniectomy due to refractory intracranial hypertension, etc) is determined by attending neurosurgeon.

CONTACTS AND LOCATIONS:
Overall Officials: Jinfang Liu, M.D., Principal Investigator — Xiangya Hospital of Central South University

IPD SHARING:
Plan to Share IPD: No